CLINICAL TRIAL: NCT04687280
Title: Comparison of Multiphase and Monophasic Arterial Hepatic MRI in the Detection of Arterial Enhancement of CHC Nodules in Cirrhotic Patients
Brief Title: Comparison of Multiphase and Monophasic Arterial Hepatic MRI in the Detection of Arterial Enhancement of CHC Nodules
Acronym: CHIC MultiA
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-24b
Record Dates: First submitted 2020-11-26; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional — non interventional, study on data

SUMMARY:
The detection and diagnosis of hepatocellular carcinoma is a public health issue. MRI is the most sensitive examination for diagnosis and especially hypervascularization in the arterial phase.

Several studies have shown that MRI multiphase arterial sequences are superior to single phase to capture the arterial phase. The purpose of this study is to compare arterial enhancement sensibilities between multi and single phase sequences.

ELIGIBILITY:
Inclusion Criteria:

* patient included in CHIC study with histology of hepatocellular carcinoma

Exclusion Criteria:

* nodules already treated by chimioembolization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient followed up for cirrhosis with discovery of a suspicious CHC nodule during imaging monitoring
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2009-04-22 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
arterial enhancement | 1 year
  significant arterial enhancement present in one of the three phases of multiphasic arterial time compared to all other arterial phases or single phase